CLINICAL TRIAL: NCT05175755
Title: Genetic Risk Factors Predictive of the Occurrence of Maternally Diagnosed Perinatal Depression in Women
Acronym: PsyCOVIDUMGEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PsyCOVIDUMGEN
Record Dates: First submitted 2021-12-30; First posted 2022-01-04 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-02

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): The procedure involves taking a total of 12 ml of blood.
  Interventions: Other: Patients

INTERVENTIONS:
Other: Patients — The procedure involves taking a total of 12 ml of blood.

SUMMARY:
In December 2019, infection with a novel coronavirus SARS-CoV-2 emerged in China and has since spread throughout the world. Forms of varying severity of COVID-19, a disease induced by this emerging virus, have been described in pregnant women. In addition to the direct effects of the virus on the pregnant woman and the fetus, the pandemic context itself is likely to act as a psychological risk factor and to alter the protective factors for mental disorders. This pandemic context is in itself anxiety-provoking, even traumatogenic, particularly because of the potentially lethal infectious risk that it carries, all the more so in psychologically vulnerable populations. In addition to the fear of viral contamination, in the perinatal period, the fear of childbirth also includes a more or less important part of anxiety-producing uncertainty. This addition of stress factors is likely to increase the prevalence of perinatal anxiety disorders, particularly psychotraumatic experiences of childbirth and peri-traumatic dissociative states. Health and social measures, such as confinement, restriction of access of accompanying persons to maternity services, or contagious isolation of mothers suspected of being infected or infected, which may furthermore impose a mother-infant separation, are also likely to have psychopathological consequences.

Studies specifically concerning the psychological effects of the COVID-19 pandemic context have been published. Among them, the French COVIPREV study, carried out in the general population during the first and second week of the containment period (beginning mid-March 2020), reported a prevalence of anxiety of 26.7% and 21.5% respectively. These prevalences are significantly higher than the usual prevalence estimated at 13.5% in the same population. Many international studies show an increase in the prevalence of postnatal depression in the current pandemic context. In the population of pregnant women, an Italian study on the psychological impact of the COVID-19 pandemic in 100 women in pregnancy, with no psychiatric history, in Naples during the second half of March 2020, found a positive score on the Impact of Event Scale-Revised (IES-R) for more than half of the women and a positive anxiety score on the State-Trait Anxiety Inventory (STAI-S) for 68% of the women The same observation was made in Quebec where two cohorts of pregnant women (between 4 and 41 weeks of amenorrhea) subjected to self-questionnaires evaluating different dimensions of their mental health, a first one recruited before the pandemic phase of 496 women and a second one of 1258 women recruited online between April 2 and 13, 2020, have been analyzed. Women in the second cohort had significantly higher levels of depressive and anxiety symptoms, more dissociative symptoms and post-traumatic stress symptoms. In China, a multicenter study in 25 hospitals in 10 provinces across the country that included 4124 women in the third trimester of pregnancy from January 1 to February 9, 2020, when the epidemic was publicly announced on January 20, 2020, again reported increased levels of anxiety and depressive symptoms on the Edinburgh Postnatal Depression Scale (EPDS) in pregnant women after the announcement compared to before. Finally, similar results are reported by Turkish researchers showing again a high prevalence of depressive symptoms during pregnancy (35.4%) during the COVID-19 pandemic. In the perinatal context, it has been documented that post-traumatic stress disorder is strongly associated with the risk of perinatal depression.

In the context of the COVID-19 pandemic, three maternity units of the PREMA University Hospital Federation (FHU PREMA), the Paris Saint-Joseph Hospital Group (GhPSJ), the Louis Mourier Hospital (APHP) and the Port-Royal Maternity Unit (APHP), in partnership with the Boulevard Brune Psychopathology Center (CPBB) and the Psychiatry Department of the Louis Mourier Hospital (APHP), have set up, as of June 2020 a care protocol consisting of a screening offered systematically to women in postpartum at D1 of their delivery, intended to identify those presenting anxiety and depressive perinatal symptoms using the Edinburgh Postnatal Depression Scale (EPDS). Thus, the PsyCOVIDUM project to estimate the prevalence of depressive symptoms in the immediate postpartum period just after delivery at different times during the pandemic episode was initiated in the three FHU PREMA maternity hospitals.

This study aims at the constitution of a DNA and serum biobank in voluntary women presenting or not a depression with an antenatal onset identified at the maternity hospital. This collection would eventually allow the evaluation of the role of inflammatory and genetic biological factors in the occurrence of antenatal onset depression on an independent cohort.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman whose age is ≥ 18 years, delivering after 34 SA in one of the two participating maternity hospitals that responded to the EPDS
* Accepting a blood sample
* EPDS score less than 8 or greater than 11
* French-speaking woman
* Woman affiliated with a health insurance plan
* Free, informed, written consent was obtained from the woman

Exclusion Criteria:

* Fetal death or medical termination of pregnancy
* Women under guardianship or trusteeship
* Woman deprived of liberty
* Woman under court protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Role of genetic factors involved in maternally diagnosed perinatal depression by genome-wide association analysis | Day 3
  This outcome corresponds to the biobank built up from the blood samples of the included female volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Elie AZRIA, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Maternité Louis Mourier, Colombes
  - Groupe Hospitalier Paris Saint-Joseph, Paris

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Chen H, Guo J, Wang C, Luo F, Yu X, Zhang W, Li J, Zhao D, Xu D, Gong Q, Liao J, Yang H, Hou W, Zhang Y. Clinical characteristics and intrauterine vertical transmission potential of COVID-19 infection in nine pregnant women: a retrospective review of medical records. Lancet. 2020 Mar 7;395(10226):809-815. doi: 10.1016/S0140-6736(20)30360-3. Epub 2020 Feb 12. PMID 32151335
- [Background] Kayem G, Lecarpentier E, Deruelle P, Bretelle F, Azria E, Blanc J, Bohec C, Bornes M, Ceccaldi PF, Chalet Y, Chauleur C, Cordier AG, Desbriere R, Doret M, Dreyfus M, Driessen M, Fermaut M, Gallot D, Garabedian C, Huissoud C, Luton D, Morel O, Perrotin F, Picone O, Rozenberg P, Sentilhes L, Sroussi J, Vayssiere C, Verspyck E, Vivanti AJ, Winer N, Alessandrini V, Schmitz T. A snapshot of the Covid-19 pandemic among pregnant women in France. J Gynecol Obstet Hum Reprod. 2020 Sep;49(7):101826. doi: 10.1016/j.jogoh.2020.101826. Epub 2020 Jun 4. PMID 32505805
- [Background] Rasmussen SA, Jamieson DJ. Coronavirus Disease 2019 (COVID-19) and Pregnancy: Responding to a Rapidly Evolving Situation. Obstet Gynecol. 2020 May;135(5):999-1002. doi: 10.1097/AOG.0000000000003873. PMID 32213786
- [Background] Walker KF, O'Donoghue K, Grace N, Dorling J, Comeau JL, Li W, Thornton JG. Maternal transmission of SARS-COV-2 to the neonate, and possible routes for such transmission: a systematic review and critical analysis. BJOG. 2020 Oct;127(11):1324-1336. doi: 10.1111/1471-0528.16362. Epub 2020 Jul 22. PMID 32531146
- [Background] Shigemura J, Ursano RJ, Morganstein JC, Kurosawa M, Benedek DM. Public responses to the novel 2019 coronavirus (2019-nCoV) in Japan: Mental health consequences and target populations. Psychiatry Clin Neurosci. 2020 Apr;74(4):281-282. doi: 10.1111/pcn.12988. Epub 2020 Feb 23. No abstract available. PMID 32034840
- [Background] Achtyes E, Keaton SA, Smart L, Burmeister AR, Heilman PL, Krzyzanowski S, Nagalla M, Guillemin GJ, Escobar Galvis ML, Lim CK, Muzik M, Postolache TT, Leach R, Brundin L. Inflammation and kynurenine pathway dysregulation in post-partum women with severe and suicidal depression. Brain Behav Immun. 2020 Jan;83:239-247. doi: 10.1016/j.bbi.2019.10.017. Epub 2019 Nov 5. PMID 31698012